CLINICAL TRIAL: NCT02972931
Title: Impact of Antiretroviral Treatment and Predictors in Subjects With Extremely Low HIV-1 Reservoir: Optimization of New Cure Strategies
Brief Title: LoViReT (Low Viral Reservoir Treated Patients)
Acronym: LoViReT
Status: Completed | Type: Observational
Sponsor: IrsiCaixa (Other)
Responsible Party: Sponsor
Other Study IDs: LoViReT
Record Dates: First submitted 2016-11-17; First posted 2016-11-25 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-10

CONDITIONS: Hiv
Keywords: HIV infection; low HIV reservoir; functional cure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LoViReT: HIV-infected subjects with extremely low or undetectable HIV-1 DNA levels in peripheral blood despite having initiated cART during chronic HIV-1 infection
- Standard Reservoir Level: HIV-infected subjects who initiated cART during chronic HIV-1 infection and that show standard HIV-1 DNA levels in peripheral blood

SUMMARY:
The main purpose of this study is to unravel the mechanisms by which the "Low Viral Reservoir Treated" patients (LoViReT) maintain extremely low HIV-1 DNA levels despite having initiated cART during chronic HIV-1 infection. This group may have specific and different clinical, virological and immunogenetical characteristics, compared to patients with regular reservoir size, which might be useful to design new and more effective treatment approaches.

DETAILED DESCRIPTION:
Combination antiretroviral therapy (cART) is highly successful suppressing HIV-1 replication and clinical progression in infected patients. However, it does not hamper the establishment of viral reservoirs, generating latently infected cells that provoke a quick rebound of HIV viremia after treatment interruption. Different strategies to tackle HIV-1 reservoirs have been suggested during last years with limited success. Actually, the few cases of described HIV-1 functional cure are found in elite and post-treatment controllers. Thus, some patients with regular HIV progression can control replication spontaneously, most of them after receiving cART during primary HIV-1 infection. Indeed, the "Mississippi baby", who was treated 36h after birth, had sustained undetectable viremia for 27 months after treatment interruption. Recently, it has also been proven in successfully treated patients that low proviral reservoir is related to better HIV-1 control after treatment discontinuation. Thus, the identification of patients with lower latent reservoir in chronic infection will allow unveiling potential mechanisms to achieve a functional cure after cART withdrawal.

Our center in Badalona allocates a biological sample collection containing 72,000 specimens from HIV-1-infected subjects. Samples from 319 patients under suppressive cART for more than 3 years have been screened using the high sensitive BioRad droplet digital Polymerase Chain Reaction platform (ddPCR). Among the screened patients, a cohort of 20 "Low Viral Reservoir Treated" patients (LoViReT) with extremely low or undetectable HIV-1 DNA levels in peripheral blood despite having initiated cART during chronic HIV-1 infection have been established, which is expected to be increased up to 40 patients. Discovering the factors that reduce HIV reservoir and make LoViReT patients maintain extremely low levels of proviral HIV-1 DNA will open new treatment strategies based on maintaining the reservoir to the lowest levels beside the regular clinical marker of viral load. In addition, a further second step of controlled cART interruption can be designed to evaluate the real impact of harboring extremely low levels of latent reservoir for further functional HIV cure.

To unravel the mechanisms by which the LoViReT cohort maintain extremely low HIV-1 DNA levels despite having initiated cART during chronic HIV-1 infection, this cohort will be studied from different points of view. All the results will be compared to a control group of 40 individuals with standard levels of total HIV DNA (reservoir). Three mayor aims will be addressed to then extrapolate our results to larger chronic HIV-1-infected populations:

* To investigate the role of cART on the suppression of the HIV reservoir in the LoViReT patients, compared to controls. To address this objective, a longitudinal analysis of proviral HIV DNA for each patient will be performed, including time points previous to cART. In total, 200 samples will be analyzed and dynamic models will be built for the two different levels of reservoir establishment. General immune phenotype of cellular populations, including also activation markers, will be also assessed in all time points.
* To investigate the integrity of HIV sequences in the LoViReT patients and its relationship with pathogenesis, in comparison to controls. Genotypic HIV tropism and the full viral genome will be analyzed through sequencing from DNA of patients' Peripheral Blood Mononuclear Cells (PBMC). Fresh blood samples will be taken from the 40 LoViReT and 40 control patients in the study. In addition, for those exerting virus production, viral isolates will be used to analyze viral replication capacity and cell pathogenesis.
* To investigate the role of immune-genetic factors that along with cART contribute to reduce the HIV reservoirs in the LoViReT patients. Functional T-cell response will be measured isolating CD8 T cells and measuring the inhibition capacity for HIV replication in each patient. Specific HIV-related CD8 T-cell interferon production will be also evaluated under epitope stimulus. Other progression associated genetic factors as Human Leukocyte Antigen (HLA) type, and chemokine receptor 5 (CCR5) and 2 (CCR2), and SIGLEC-1 Single Nucleotide Polymorphisms (SNPs) will be also explored.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Voluntarily signed informed consent
* Proven HIV-1 infection
* On stable cART regimen (antiretroviral therapy consisting of at least 3 registered antiretroviral agents) for at least 3 years
* HIV-RNA <50 copies/mL during the last 3 years prior to the study
* Proviral HIV-DNA <50 copies/million PBMCs by using the ultrasensitive BioRad residual ddPCR quantification platform

Exclusion Criteria:

* cART discontinuation between previous screening and Visit #1.
* HIV-RNA above 50 copies/mL between previous screening to Visit #1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected subjects with extremely low or undetectable HIV-1 DNA levels in peripheral blood despite having initiated cART during chronic HIV-1 infection
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martinez-Picado, PhD, Principal Investigator — IrsiCaixa AIDS Research Institute, Hospital Universitari Germans Trias i Pujol
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvez C, Urrea V, Dalmau J, Jimenez M, Clotet B, Monceaux V, Huot N, Leal L, Gonzalez-Soler V, Gonzalez-Cao M, Muller-Trutwin M, Saez-Cirion A, Garcia F, Blanco J, Martinez-Picado J, Salgado M. Extremely low viral reservoir in treated chronically HIV-1-infected individuals. EBioMedicine. 2020 Jul;57:102830. doi: 10.1016/j.ebiom.2020.102830. Epub 2020 Jun 21. PMID 32580136
- [Background] Galvez C, Urrea V, Garcia-Guerrero MDC, Bernal S, Benet S, Mothe B, Bailon L, Dalmau J, Martinez A, Nieto A, Leal L, Garcia F, Clotet B, Martinez-Picado J, Salgado M. Altered T-cell subset distribution in the viral reservoir in HIV-1-infected individuals with extremely low proviral DNA (LoViReTs). J Intern Med. 2022 Aug;292(2):308-320. doi: 10.1111/joim.13484. Epub 2022 Mar 28. PMID 35342993

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Reanalysis of total HIV DNA in 30 LoViReT and 32 control patients of the cohort was made, and 22 LoViReT patients and 22 controls were finally selected for the study (the ones still fulfilling criteria).
  In terms of apheresis and tissue samples of the LoViReT patients, we finally collected: 14 apheresis, 8 lymph node FNB and 8 rectal biopsies.
Period: Overall Study
Arm/Group | LoViReT | Standard Reservoir Level
Started | 30 | 32
Completed | 22 | 22
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LoViReT | Standard Reservoir Level | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.70 [44.14 to 53.84] | 51.01 [46.90 to 58.11] | 50.70 [46.40 to 57.71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 17 | 20 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 20 | 17 | 37
  Race: Non caucasian | 0 | 5 | 5
  Race: Not available | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Analysis of Total HIV DNA and Immune-phenotype by Digital Droplet Polymerase Chain Reaction (PCR) and Flow Cytometry, Respectively, Comparing This Outcome Before and After cART (Evaluation of cART Effect on This Parameters)
Description: To address this objective, a longitudinal analysis of proviral HIV DNA for each patient will be performed, including time points previous to cART. In total, 200 samples will be analyzed and dynamic models will be built for the two different levels of reservoir establishment. General immune phenotype of cellular populations, including also activation markers, will be also assessed in all time points.
Time Frame: The time frame for the outcome measure is an average of 5 years. Including a baseline, 18 months, and 5 years post cART initiation.
Population: The participants analyzed correspond to a subgroup of participants with sample availability for all the timepoints analyzed, and started cART during chronic HIV-1 infection.
Measure: Median (Inter-Quartile Range); unit: DNA copies/milion of CD4 T cells
Arm/Group | LoViReT | Standard Reservoir Level
Number analyzed (Participants) | 12 | 13
DNA copies/milion of CD4 T cells
  Baseline | 812 [485 to 1392] | 5062 [2649 to 8943]
  Last sample | 54 [38 to 67] | 714 [517 to 1462]

2. Primary Outcome: Replication Competent Reservoir in Patients With Low (LoViReT) Normal (Controls) Levels of Total HIV DNA
Description: Replication competent reservoir will be analyzed with the gold standard quantitative viral outgrowth assay (qVOA).
Time Frame: The time frame for the outcome measure is on patients on cART for at least 5 years.
Population: The participants analyzed correspond to a subgroup LoVireT who agreed to have a phlebotomy. No results for control group because de phlebotomy was not indicated.
Measure: Count of Participants; unit: Participants
Groups:
- Loviret: HIV-infected subjects with extremely low or undetectable HIV-1 DNA levels in peripheral blood
Arm/Group | Loviret
Number analyzed (Participants) | 14
Participants
  Positive | 4
  Negative | 10

3. Primary Outcome: Evaluation and Comparison of CD8 T-cell Responses by Inhibition Assays, Between Patients With Low (LoViReT) and Normal (Controls) Levels of Total HIV DNA
Description: Functional T-cell response will be measured isolating CD8 T and Nk cells and measuring the inhibition capacity for HIV replication in each patient.
Time Frame: The time frame for the outcome measure is on samples before initiation of cART and after 5 years on cART
Population: 11 LoViReT and 11 controls with available samples before initiation of cART and after 5 years on cART were analyzed
Measure: Median (Inter-Quartile Range); unit: percentage of inhibition
Arm/Group | LoViReT | Standard Reservoir Level
Number analyzed (Participants) | 11 | 11
percentage of inhibition
  NK cells pre cART | 57.52 [14.54 to 77.36] | 50.17 [10.56 to 69.53]
  NK cells 5 years on cART | 38.61 [5.71 to 54.2] | 42.77 [0.88 to 63.51]
  CD8 T cells pre cART | 27.05 [0 to 39.37] | 57.33 [52.77 to 81.36]
  CD8 T cells 5 years on cART | 28.09 [0 to 57.05] | 41.21 [0 to 76.25]

4. Primary Outcome: Analysis and Comparison of Progression-associated Genetic Factors, Between Patients With Low (LoViReT) and Normal (Controls) Levels of Total HIV DNA
Description: Different progression-associated genetic factors, such as HLA type, and CCR5, CCR2 and SIGLEC-1 single nucleotide polymorphisms (SNPs) will be also explored.
Time Frame: The time frame for the outcome measure is on patients on cART for at least 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | LoViReT | Standard Reservoir Level
Number analyzed (Participants) | 22 | 22
Participants
  CCR5 genotype: wild type homozygous | 16 | 11
  CCR5 genotype: heterozygous | 6 | 3
  CCR5 genotype: mutated homozygous | 0 | 0
  CCR5 genotype: Not available | 0 | 8
  Siglec-1 genotype: wild type homozygous | 21 | 21
  Siglec-1 genotype: heterozygous | 1 | 1
  Siglec-1 genotype: mutated homozygous | 0 | 0
  Siglec-1 genotype: Not available | 0 | 0

5. Primary Outcome: Measurement of Genotypic Tropism in Patients With Low (LoViReT) and Normal (Controls) Levels of Total HIV DNA
Description: Genotypic HIV tropism and the full viral genome will be analyzed through sequencing from DNA of patients' peripheral blood mononuclear cells (PBMC).
Time Frame: The time frame for the outcome measure is on patients on cART for at least 5 years.
Population: Loviret and controls were analyzed for virus tropism
Measure: Count of Participants; unit: Participants
Groups:
- Control: HIV-infected subjects who initiated cART during chronic HIV-1 infection and that show standard HIV-1 DNA levels in peripheral blood
Arm/Group | Loviret | Control
Number analyzed (Participants) | 22 | 22
Participants
  CCR5 | 12 | 18
  CXCR4 | 1 | 3
  Not determined | 9 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: The clinical investigators were responsible for detecting and documenting any event that meets the criteria and definitions of adverse event (AE) or serious adverse event (SAE) for this protocol.
  Adverse events occurred during the visit were recorded in the database and included in the final report.
Arm/Group | LoViReT | Standard Reservoir Level
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LoViReT (N=22) | Standard Reservoir Level (N=22)
Saddle dermatoma (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LoViReT (N=22) | Standard Reservoir Level (N=22)
Swelling (General disorders) | 2 (2) | 0 (0)
Acute bronchitis (Infections and infestations) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
As expected and included in the protocol, not all participants were willing to provide all the types of samples, but relevant results were obtained anyway.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02972931/Prot_SAP_000.pdf